CLINICAL TRIAL: NCT04553328
Title: Ultrasound-guided Ipsilateral Transverse Abdominis Plane and Ilioinguinal-iliohypogastric Nerve Block Versus Ipsilateral Illioinguinal- Illiohypogastric Nerve Block for Inguinal Hernia Repair in Patients With Liver Cirrhosis
Brief Title: Ultrasound-guided Ipsilateral Transverse Abdominis Plane and Ilioinguinal Iliohypogastric Nerve Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Salah Eldin Mahmoud Badre, Clinical Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU R 48/2019
Record Dates: First submitted 2020-08-14; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Liver Cirrhosis
Keywords: Transverse aabdominis plane
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: The patients were divided randomly into two groups (30 patients in each group) according to the type of block they received: Group (T) received ultrasound guided (US) combined ipsilateral transverse abdominis plane (TAB) and ilioinguinal- iliohypogastric (ILIH) nerve block. Group (I) received US guided ipsilateral illioinguinal- illiohypogastric nerve block only.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): Group (T) received ultrasound guided (US) combined ipsilateral transverse abdominis plane (TAB) and ilioinguinal- iliohypogastric (ILIH) nerve block
  Interventions: Device: Us guided nerve blocks
- Group I (Active Comparator): Group (I) received US guided ipsilateral illioinguinal- illiohypogastric nerve block only.
  Interventions: Device: Us guided nerve blocks

INTERVENTIONS:
Device: Us guided nerve blocks — The ILIH nerves were identified and located in the fascia compartment between the internal oblique and the transverse abdominis or external oblique muscles, a 20 G needle was advanced between the aponeurosis of the internal oblique and transverses abdominis muscles then 30 ml bupivacaine 0.25% was injected with intermittent aspiration,then 10 ml bupivacaine 0.25% was injected around the nerves.
  Other Names: drug used is bupivacaine

SUMMARY:
The purpose of this study is to compare the efficacy of using TAB and ILIH nerve blocks versus ILIH nerve block only for inguinal hernia repair in patients with liver cirrhosis.

DETAILED DESCRIPTION:
After obtaining institutional ethical committee approval and written informed consent in 2019, 60 patients between the age of 40 and 70 year were divided randomly using a computer generated randomization table and opaque sealed envelopes into two groups (30 patients in each group) according to the type of block they received: Group (T) received ultrasound guided (US) combined ipsilateral transverse abdominis plane (TAB) and ilioinguinal- iliohypogastric (ILIH) nerve block. Group (I) received US guided ipsilateral illioinguinal- illiohypogastric nerve block only.

Standard monitoring was used throughout the surgery; heart rate (HR), non-invasive mean arterial blood pressure (MAP), respiratory rate (RR) and oxygen saturation (SpO2)documented at baseline before the block then at 5-min intervals intraoperative , then during the immediate postoperative period at 15 and 30 min, and at discharge from the PACU.

A nasal prong was applied and supplemental oxygen at 3 l/min of fresh gas flow was given throughout the procedure. It was explained clearly to the patients that any pain, discomfort, or anxiety would be managed by the administration of local anesthetic (LA) infiltration with bupivacaine 0.25% during the operation or by conversion to general anesthesia (GA) if needed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification groups II and III,undergoing unilateral inguinal hernia repair.
* All patients have liver cirrhosis having a Child-Pugh classification of liver disease (3) class B with a score ≤ 8/15,
* Moemen modified classification of liver disease (4) class B,
* an international normalized ratio (INR)≤1.5.

Exclusion Criteria:

* Patients with Child-Pugh ≥ 8/15,
* INR≥ 1.5,
* Grade 3 ascites,
* Serum sodium ≤120 meq/l,
* Recurrent hernia, or bilateral hernia,
* Body mass index (BMI) ≥ to 40 kg/m 2,
* known allergy to any of the medicines used
* Any renal or cardiovascular dysfunction, bronchial asthma, hematological disorders (other than secondary to chronic liver disease),
* Patient refusal.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
local anesthetic infiltration and convesion to general anesthesia | data will be reported and assessed within 24 weeks.
  need for additional local anesthetic infiltration and conversion to general anesesthesia by assessing sensory block adequacy with thermal sensation using an alcohol swab.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Badre, PHD, Principal Investigator — Associate professor of Anesthesia and ICU, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Final results are to be shared with other researchers after approval of publication
Supporting Information: Study Protocol
Time Frame: within 1 month , for 3 years
Access Criteria: anesthesia doctors in same field